CLINICAL TRIAL: NCT05496543
Title: A Randomized Controlled Clinical Trial of Acupuncture in Nourishing Kidney and Dredging Fu Organs for Functional Constipation in Older Adults
Brief Title: Acupuncture for Functional Constipation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yin Ping (Other)
Collaborators: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Longhua Hospital (Other)
Responsible Party: Sponsor-Investigator, Yin Ping, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21Y11923900
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Participants will receive acupuncture treatment at Zhao Hai(KI 6), Da Zhong(KI 4), Tai Xi(KI 3), Tian Shu(ST 25), and Shang Ju Xu(ST 37) bilaterally.
  Each treatment will last 30 minutes and participants will receive the treatment 3 times per week (every other day) for 8 weeks, 24 sessions in total. Follow-up time is week 4 and week 12 after treatment (ie, week 12 and week 20).
  Interventions: Device: acupuncture
- Sham acupuncture group (Placebo Comparator): Participants will receive sham acupuncture treatment on bilateral sham Zhao Hai(KI 6), Da Zhong(KI 4), Tai Xi(KI 3), Tian Shu(ST 25), and Shang Ju Xu(ST 37) that match real acupuncture points.
  The duration of needle retention, treatment period, and follow-up in the control group is the same as that in the intervention group.
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: acupuncture — All acupoints will be routinely sterilized at first. After the insertion of the needles, manipulations of lifting, twirling, and thrusting are performed on all needles to reach de qi, which is a sensation typically associated with needling including soreness, numbness, swelling, heaviness, and other feelings. This is considered to be an important component of the therapeutic effect of acupuncture.
  Arms: Acupuncture group
Device: sham acupuncture — The placebo needles chosen for this study are flat-tipped needles without a tip, which could not be pierced into the skin. In the meanwhile, an external patch device will fix the needles, which are visually pierced into the skin. After the treatment, the acupuncturist will press the acupuncture point with a dry cotton ball so that the patient can feel the pulling out of the "needle".
  Arms: Sham acupuncture group

SUMMARY:
Through a scientific and standardized randomized controlled study, we observe the effectiveness and safety of acupuncture in the treatment of functional constipation in the elderly through the method of "nourishing kidney and dredging Fu organs".

DETAILED DESCRIPTION:
Functional constipation is a common disease of old people. To date, there has not specific therapy on it. Former research showed acupuncture may work for functional constipation. In the trial, patients in the acupuncture and sham acupuncture groups will receive 24 acupuncture treatments over an 8-week period. This RCT is designed to confirm the efficacy and safety of acupuncture in functional constipation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome IV Diagnostic Criteria for Constipation and TCM Diagnostic Criteria of constipation with yin deficiency syndrome;
* No gender restriction, age 60-80;
* FC that is classified as mild or moderate;
* Have not used any medicine for constipation at least 2 weeks before treatment (except emergency treatment);
* Have not participated in other medical clinical trials over the past one month;
* Those who can understand various evaluation scales, complete the evaluation and cooperate with the completion of the planned course of treatment;
* Sign the informed consent.

Exclusion Criteria:

* Irritable bowel syndrome and constipation caused by tumors, inflammatory reactions, endocrine and metabolic diseases, and drugs;
* Constipation caused by organic diseases;
* Patients with serious primary diseases such as heart, brain, liver, kidney and hematopoietic system, infectious diseases, tumors, and mental diseases;
* Those who voluntarily give up or cannot cooperate with treatment and observation due to various circumstances;
* Patients with cognitive impairment or aphasia;
* Those who take other drugs during treatment, which affect the efficacy and judgment (except emergency treatment).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The change in the mean number of CSBMs per week compared to baseline during the 8-week treatment period | At baseline, week 4 (in treatment), week 8 (end of treatment), and the follow-up period (week 12 and week 20 after randomization).
  Complete Spontaneous Bowel Movements (CSBMs) refers to the frequency of a bowel movement that occurred in the absence of laxatives or manipulation.

SECONDARY OUTCOMES:
Bristol Stool Scale | At baseline and at week 8 (end of treatment).
  A scale to classify the patient's voluntary bowel movement stool.
Patient Assessment of Constipation-Symptoms (PAC-SYM) | At baseline and at week 8 (end of treatment).
  A scale to assess the condition of the patient's constipation-related symptoms
Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) | At baseline and at week 8 (end of treatment).
  A brief but comprehensive assessment of the daily life quality of patients with FC, containing 28 items
Self-rating Anxiety Scale（SAS） | At baseline and at week 8 (end of treatment).
  A measure of somatic symptoms associated with anxiety reactions.
Self-rating Depression Scale（SDS） | At baseline and at week 8 (end of treatment).
  A self-rating scale to assess patients' depression
Weekly usage of emergency bowel medications | At baseline and at week 8 (end of treatment).
  The proportions of participants using medications and doses for emergency treatment
Incidence of adverse events | During 1-8 weeks
  The adverse events (AEs) assessment aims at evaluating the AEs of acupuncture treatment.

CONTACTS AND LOCATIONS:
Overall Officials: PING YIN, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou K, Fang J, Wang X, Wang Y, Hong Y, Liu J, Wang L, Xue C, Wang P, Liu B, Zhu B. Characterization of de qi with electroacupuncture at acupoints with different properties. J Altern Complement Med. 2011 Nov;17(11):1007-13. doi: 10.1089/acm.2010.0652. Epub 2011 Oct 14. PMID 21999154
- [Background] Dunstan DA, Scott N. Norms for Zung's Self-rating Anxiety Scale. BMC Psychiatry. 2020 Feb 28;20(1):90. doi: 10.1186/s12888-019-2427-6. PMID 32111187
- [Background] Dunstan DA, Scott N. Clarification of the cut-off score for Zung's self-rating depression scale. BMC Psychiatry. 2019 Jun 11;19(1):177. doi: 10.1186/s12888-019-2161-0. PMID 31185948